CLINICAL TRIAL: NCT04492345
Title: Impact of Isocinetism on the Disorders of the Spinal Statics of the Parkinsonian Patient
Brief Title: Assessment of a Special Modality of Back Muscles Strengthening for Postural Deformations in Parkinsonian Patient
Acronym: ISOPARK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18_RIPH2-10
Record Dates: First submitted 2020-04-21; First posted 2020-07-30 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Parkinson Disease; Physical Medicine; Rehabilitation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patient with conventional rehabilitation session and isokinetic reeducation during 7 weeks
  Interventions: Other: Isokinetic reeducation
- Control (Other): Patient with conventional rehabilitation session during 7 weeks
  Interventions: Other: Conventional reeducation

INTERVENTIONS:
Other: Isokinetic reeducation — Conventional rehabilitation session and isokinetic during 7 weeks
  Arms: Experimental
Other: Conventional reeducation — Conventional rehabilitation session during 7 weeks
  Arms: Control

SUMMARY:
Parkinson's patients have postural disorders. These disorders are frequent in Martinique. Physiotherapeutic rehabilitation is essential because these disorders are generally non dopa-sensitive.

DETAILED DESCRIPTION:
Postural disorders are very common in Martinique, in patients often having an atypical form of the Parkinson's disease. Physiotherapy rehabilitation is essential because these disorders are generally non-dopa-sensitive. Isokinetic muscle strength may reduce postural disorder in Parkinson's disease.

Isokinetic device rehabilitation promotes maximum muscular contraction at constant speed; the resistance of the machine continuously adapting to the force developed by the subject. As the spinal muscle strength gain is superior to conventional post-rehabilitation motor function, the improvement in postural instability should be greater than that achieved with conventional rehabilitation. A better postural support should thus result in a decrease in the risk of falling and an improvement in the quality of walking.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Parkinson's disease or atypical parkinsonian syndrome
* Age ≥18 years
* Patient with postural disorders with a cervical arrow> 6cm in the sagittal plane and / or the axis C7S2 different from 0 in the frontal plane
* UPDRS between 10 and 25/108.
* Antiparkinsonian treatment stabilized for 8 weeks
* MMS test> 25
* Insured person or beneficiary of social security

Exclusion Criteria:

* Patient with a neurological condition other than parkinsonian syndrome
* Patient with rheumatic disease
* Patient with a history of trunk surgery
* Patient with a brain stimulator
* Cardiac pathology not stabilized
* Incapacitated adult, or under guardianship, or under curatorship or under judicial protection curatorship

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Patient posture | After 8 weeks of reeducation
  Measure in centimetres from the arrow to C7

SECONDARY OUTCOMES:
Spinal muscle strength | After 8 weeks of reeducation
  Static contraction measured in holding time in seconds
Spinal muscle strength | After 8 weeks of reeducation
  Isokinetic contraction measured by a force in Newton/Kg and an abdominal spinal ratio of 66%.
Improvement of balance | After 8 weeks of reeducation
  Increasing the score on the BERG BALANCE SCALE BETWEEN 0 - 56.
Walking speed | After 8 weeks of reeducation
  Carry out a 10-metre Walk Test

CONTACTS AND LOCATIONS:
Overall Officials: Sabine SOPHIA, Principal Investigator — CHU Martinique
Locations (1):
- CHU de Martinique, Le Lamentin, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tiffreau V, Preudhomme M, Defebvre L. Troubles de la statique au cours des affections neurologiques évolutives: syndromes parkinsoniens et pathologies musculaires. Revue du rhumatisme monographies 78 (2011) 26-31
- [Background] Hubble RP, Naughton GA, Silburn PA, Cole MH. Trunk muscle exercises as a means of improving postural stability in people with Parkinson's disease: a protocol for a randomised controlled trial. BMJ Open. 2014 Dec 31;4(12):e006095. doi: 10.1136/bmjopen-2014-006095. PMID 25552609
- [Background] Hutin E et al, Communications orales- Maladie de Parkinson. Effet d'une kinésithérapie standardisée sur la stabilité posturale dans la maladie de Parkinson au stade modéré. CO36-002-f. Annals of Physical and Rehabilitation Medicine 56S (2013) e190-e196.
- [Background] Crizzle AM, Newhouse IJ. Is physical exercise beneficial for persons with Parkinson's disease? Clin J Sport Med. 2006 Sep;16(5):422-5. doi: 10.1097/01.jsm.0000244612.55550.7d. PMID 17016120
- [Background] Frazzitta G, Ferrazzoli D, Maestri R, Rovescala R, Guaglio G, Bera R, Volpe D, Pezzoli G. Differences in muscle strength in parkinsonian patients affected on the right and left side. PLoS One. 2015 Mar 25;10(3):e0121251. doi: 10.1371/journal.pone.0121251. eCollection 2015. PMID 25806509
- [Background] Edouard P, Degache F. Guide d'isocinétisme, L'évaluation isocinétique des concepts aux conditions sportives et pathologiques. Elsevier Masson;09/2016.
- [Background] Lannuzel A, Edragas R, Lackmy A, Tressieres B, Pelonde V, Kaptue MEN, Mecharles S, Demas A, Francois B, McGovern E, Vidailhet M, Gaymard B, Roze E. Further evidence for a distinctive atypical degenerative parkinsonism in the Caribbean: A new cluster in the French West Indian Island of Martinique. J Neurol Sci. 2018 May 15;388:214-219. doi: 10.1016/j.jns.2018.02.019. Epub 2018 Feb 6. PMID 29525296
- [Background] DiFrancisco-Donoghue J, Jung MK, Geisel P, Werner WG. Learning effects of the sensory organization test as a measure of postural control and balance in Parkinson's disease. Parkinsonism Relat Disord. 2015 Aug;21(8):858-61. doi: 10.1016/j.parkreldis.2015.05.007. Epub 2015 May 14. PMID 25997862
- [Background] Lima LO, Cardoso F, Teixeira-Salmela LF, Rodrigues-de-Paula F. Work and power reduced in L-dopa naive patients in the early-stages of Parkinson's disease. Arq Neuropsiquiatr. 2016 Apr;74(4):287-92. doi: 10.1590/0004-282X20160014. PMID 27097000
- [Background] Durmus B, Baysal O, Altinayar S, Altay Z, Ersoy Y, Ozcan C. Lower extremity isokinetic muscle strength in patients with Parkinson's disease. J Clin Neurosci. 2010 Jul;17(7):893-6. doi: 10.1016/j.jocn.2009.11.014. PMID 20435478
- [Background] Cano-de-la-Cuerda R, Vela-Desojo L, Miangolarra-Page JC, Macias-Macias Y. Isokinetic dynamometry as a technologic assessment tool for trunk rigidity in Parkinson's disease patients. NeuroRehabilitation. 2014;35(3):493-501. doi: 10.3233/NRE-141142. PMID 25260231
- [Background] Gracies JM. [Neurorehabilitation in parkinsonian syndromes]. Rev Neurol (Paris). 2010 Feb;166(2):196-212. doi: 10.1016/j.neurol.2009.10.026. Epub 2010 Feb 6. French. PMID 20138321
- [Background] Tambosco L et al, Communications orales- Maladie de Parkinson. Particularités de la réponse à l'effort chez les patients atteints d'une maladie de Parkinson. CO36-003-f. Annals of Physical and Rehabilitation Medicine 56S (2013) e190-e196.
- See also: Isocinetique_easytech_guide_clinique.pdf — https://www.elitemedicale.fr/genu-plus-easytech